CLINICAL TRIAL: NCT04552613
Title: Efficacy of Targeted Therapy Combined Chemotherapy in Advanced EGFR Positive NSCLC Patients With Concurrent Driver Gene Mutations
Brief Title: Efficacy of Targeted Therapy Combined Chemotherapy in Advanced EGFR Positive NSCLC Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K2020109
Record Dates: First submitted 2020-09-13; First posted 2020-09-17 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Non-small-lung-cell Cancer; NSCLC; EGFR Gene Mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard programme group (Experimental): EGFR-TKI targeted therapy
  Interventions: Drug: EGFR-TKI
- controlled programme group (Active Comparator): EGFR-TKI targeted therapy combined chemotherapy(pemetrexed plus carboplatin for 4 cycles )
  Interventions: Drug: EGFR-TKI combined with chemotherapy (pemetrexed plus carboplatin)

INTERVENTIONS:
Drug: EGFR-TKI — (A) Standard programme group, EGFR-TKI targeted therapy;
  Arms: Standard programme group
Drug: EGFR-TKI combined with chemotherapy (pemetrexed plus carboplatin) — (B) controlled programme group, EGFR-TKI targeted therapy combined chemotherapy(pemetrexed plus carboplatin for 4 cycles )
  Arms: controlled programme group

SUMMARY:
This study is a randomized, multicenter clinical study ，which is designed to compare the efficacy of the safety and efficacy of treatment every 6 weeks in EGFR positive (Non-small cell lung cancer, NSCLC) with concurrent Driver gene mutations，who used EGFR-TKI with or without combined chemotherapy，estimated with stable efficacy (CR, PR, and SD) .In this study, subjects will be randomly assigned to the following two groups according to a 1:1 ratio:(A) Standard programme group, EGFR-TKI targeted therapy; (B) controlled programme group, EGFR-TKI targeted therapy combined chemotherapy(pemetrexed plus carboplatin for 4 cycles )

DETAILED DESCRIPTION:
This study is a randomized, multicenter clinical study aimed at EGFR positive non-small-cell lung cancer (NSCLC) subjects with concurrent Driver gene mutations who have not previously received systematic treatment. After comparing EGFR-TKI alone or EGFR-TKI combined with chemotherapy for 4 cycles, after the efficacy evaluation was stable (CR, PR, and SD), the safety and clinical efficacy of maintenance therapy every 6 weeks were compared. The eligible subjects in this study will be randomly assigned into the following two groups according to the 1: 1 ratio: (A) Standard programme group, EGFR-TKI targeted therapy; (B) controlled programme group, EGFR-TKI targeted therapy combined chemotherapy (pemetrexed plus carboplatin for 4 cycles ) During the course of the trial treatment, if the subject develops disease (the first PD), the researcher will decide whether to continue the medication according to the patient's situation and communicate with the patient, as follows: After the first PD of the subject, the researcher decides whether to continue the treatment with the original regimen according to the disease state of the subject. At least 4 weeks later, the tumor is evaluated again. If the tumor progresses again (the second PD), the subject's study treatment ends and the follow-up period is entered; if there is no progress, the original regimen is continued.

The primary end point was descriptive analysis of progression-free survival and Objective response rate.The secondary end point of this study was to compare the incidence of treatment-related grade 3-5 adverse events between the standard group and the controlled group. Using RECIST 1.1 as the evaluation standard, the independent imaging evaluation committee (IRRC) conducted the evaluation. For the first time to evaluate PD, regardless of whether they continue to study treatment after progression, the date of the first PD evaluated by IRRC will be used for all statistical analysis containing progress information.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer for clinical research, fully understand, inform and sign informed consent forms (Informed Consent Form, ICF), willing to follow and be able to complete all trial procedures.
2. 18 to 80 years old (with critical values) when signing ICF.
3. Histopathology or hemology diagnostics of phase IIIB or IV (AJCC Version 8) NSCLC that cannot be surgicalor-able or radiotherapy.
4. Patients have never received systemic treatment throughout the body for phase IIIB or IV NSCLC(Neoadjuvant or adjuvant chemotherapy is excluded).
5. Known EGFR sensitivity mutations with concurrent other Driver gene mutations, such as T790M，TP53，RB1，PTEN，CDKN，PIK3A，DDR, KRAS and so on.
6. The end of non-systematic anti-tumor therapy is not only 2 weeks from the end of the study drug, and the treatment-related AE is restored to CTCAE 4.03 to level 1 (except for level 2 hair loss).
7. Within 4 weeks prior to randomization, at least one measurable target lesions assessed by irRC in accordance with RECIST 1.1 requirements.
8. The ECOG PS score for 7 days prior to the first drug use of the study drug was 0 or 1.
9. The expected lifetime is more than 12 weeks.
10. The main organ function sits well, i.e. meets the following criteria (no blood transfusion, albumin, recombinant human platelet production or Colony-stimulating factor (CSF) treatment within 14 days prior to the first drug use in this study):

(1). Absolute neutrophil count >15.0 x 10^9/L; (2). Platelet count ≥ 100 x 10^9/L; (3). Hemoglobins ≥ 90 g/L; (4). Total bilirubin ≤.5 x ULN (except Gilbert syndrome, total bilirubin ≤ 3.0 mg/dL); (5). AST (SGOT) ≤ 2.5 x ULN, for patients with liver metastasis, ≤5.0 x ULN; (6). ALT (SGPT) is 2.5 x ULN, for patients with liver metastasis, ≤5.0 x ULN; (7). Clotting function: activated part of the clotting enzyme time (APTT) ≤ 1.5 x ULN, clotting enzyme raw time (PT) or international standardized ratio (INR) ≤1.5 x ULN; (8). Creatinine ≤1.5xULN, or creatinine clearance ≥60 mL/min (Cockcroft-Gault method).

11. Female patients must meet one of the following:

1. . Menopause (defined as having no menstruation for at least 1 year and no other reason for confirmation other than menopause);
2. . Sterilization performed (removal of the ovaries and/or uterus);
3. . Fertility, but must meet: Serum pregnancy tests must be negative within 7 days of randomization and agree to use 1% annual failure rate of contraception or to maintain abstinence (avoiding heterosexual intercourse) (at least 120 days after the signing of an informed consent form to the last time the drug was administered) (1% annual failure rate of contraceptive methods including bilateral tubal ligation, male sterilization, correct use of ovulation-suppressing hormones, release of intrauterine and intrauterine devices) and intrauterine devices.

12. Male patients must meet the requirement to consent to abstinence (avoiding heterosexual intercourse) or to take contraception, provided that when the partner is a woman of childbearing age or who is pregnant, male patients must maintain abstinence or use condom contraception to prevent exposure to the embryo during treatment and for at least 150 days after the end of administration of the drug. Regular abstinence (e.g. calendar days, ovulation periods, basic body temperature or late-stage contraception) and in vitro ejaculation are substandard methods of contraception.

Exclusion Criteria:

1. Received any of the following treatments: received systemic anti-tumor therapy (except neoadjuvant or adjuvant chemotherapy) previously; Within 4 weeks before the first administration of the drug, more than 30% of the bone marrow was treated with radiotherapy or a large area of radiation was carried out (except palliative radiotherapy for the purpose of relieving pain in non-target lesions only ); Other anti-tumor therapies, including molecular targeted therapies (EGFR TKI, angiogenesis inhibitors, etc.), immunotherapy (such as cellular immunotherapy anti-PD-1 or PD-L1), other experimental drug therapies, etc.
2. Major surgery was performed within 4 weeks before the first administration of the study drug.
3. Patients were taking (or cannot stop taking) certain medications or herbal supplements that are known to be a strong inducer of cytopigment P450 (CYP450) 3A4 within 1 week prior to the first administration of the study drug.
4. Patients with dysphagia or possible absorption disorders as determined by the researcher.
5. Within 5 years or at the same time, there are other active malignancies. Cured limited tumors, such as skin base cell carcinoma, skin squamous carcinoma, superficial bladder cancer, prostate in situ cancer, cervical in situ cancer, etc. can be included in the group.
6. Patients with brain metastasis, the following could except:the largest diameter of brain metastasis lesions is less than 2 cm and no obvious symptoms; brain metastatic lesions have control, and stability more than 4 weeks.
7. Resting electrocardiogram (ECG) in rhythm, conduction and morphologically abnormal clinical significance, such as complete left bundle branch block, Ⅱ degrees above heart block, PR interval period > 250 milliseconds, etc.; myocardial infarction occurred within 6 months; presence of risk factors for prolonged QT interval or increased arrhythmia, such as heart failure, moderate or severe hypokalemia, diagnosed or suspected congenital long QT syndrome, a family history of long QT syndrome, or a history of sudden death under the age of 40 in a first-degree relative; mean QT interval (QTcF) after 3 Fridericia adjustments of electrocardiogram: > 450ms for males and > 470ms for females.
8. Pregnant or lactating women.
9. Hepatitis B virus infection (HBsAg positive, HBV-DNA >1000cps/ml and AST or ALT>2.0xULN), hepatitis C virus infection or HIV infection which is not controlled or in active.
10. Other uncontrolled concomitant diseases include, but are not limited to infectious or active infections.
11. A history of epilepsy, mental illness, or other social factors that limit adherence to the program.
12. The researcher considers it inappropriate to participate in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2023-09-24 (Actual); Study Completion 2023-09-24 (Actual)

PRIMARY OUTCOMES:
progression-free survival | three years
  Patients with oncological diseases have a period of time from the start of treatment to the observation of disease progression or death due to any cause
objective response rate | three years
  Refers to the proportion of patients whose tumor shrinkage reaches a certain amount and remains for a certain period of time, including CR + PR cases

SECONDARY OUTCOMES:
overall survival | three years
  The time from randomization to death due to any cause. For subjects who have been lost to follow-up before death, the time of the last follow-up is usually calculated as the time of death.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Wang, PhD, Study Chair — The Fourth Affiliated Hospital of Zhejiang University
Locations (1):
- China, Zhejiang, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No